CLINICAL TRIAL: NCT01942954
Title: Executive Functioning in Patients With Alcohol Use Disorder Following a Mobile Health Cognitive Stimulation Approach: a Randomized Controlled Trial
Brief Title: Health Mobile Cognitive Stimulation in Alcohol Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pedro Gamito (Other)
Collaborators: Universidade Lusófona de Humanidades e Tecnologias (Other)
Responsible Party: Sponsor-Investigator, Pedro Gamito, PhD (Full Professor), Universidade Lusófona de Humanidades e Tecnologias
Organization: Universidade Lusófona de Humanidades e Tecnologias (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SLB_AUD01
Record Dates: First submitted 2013-08-30; First posted 2013-09-16 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Alcohol-Induced Disorders, Nervous System; Alcohol Dependence
Keywords: Alcohol Dependence; Cognitive Therapy; Executive Function; Mobile Health; Recovery of Function; Rehabilitation
MeSH Terms: conditions — Alcohol-Induced Disorders, Nervous System; Alcoholism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mobile health cognitive stimulation (Experimental): Experimental group
  Interventions: Other: Mobile health cognitive stimulation
- Treatment-as-usual (No Intervention): This group consists of treatment-as-usual for alcohol abstinence according to the Minnesota Model.

INTERVENTIONS:
Other: Mobile health cognitive stimulation
  Arms: Mobile health cognitive stimulation

SUMMARY:
The consequences of alcohol dependence are severe and may range from physical diseases to neuropsychological deficits in several cognitive domains. Alcohol abuse has also been related to brain dysfunction specifically in the prefrontal cortex. To assess these deficits and the application of a novel approach of cognitive stimulation to alcoholics, we have carried out a neuropsychological intervention program with mobile health technology. Patients diagnosed with alcohol dependence syndrome were submitted to cognitive stimulation during four weeks in a three-day/week basis.

ELIGIBILITY:
Inclusion Criteria:

Only patients that scored higher than the cutoff values for their age on the Mini Mental Examination Test and with no clinical scores on the Symptoms Checklist Revised were included in the study.

Exclusion Criteria:

Patients with dependency from substances other than alcohol or with history of previous neurological disorders were excluded from the study. Patients were also screened for minimal computer literacy; no patients were excluded due to lack of this criterion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-10; Primary Completion 2019-12 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Change in the results of Frontal Assessment Battery - FAB | Before cognitive rehabilitation - After cognitive rehabilitation (1month - after 10 sessions)
  The participants were assessed in Frontal Lobe Cognitive Functioning (Retention, Attention and Calculation, Language and Visual-spatial abilities)at the beginning of the rehabilitation and after 10 rehabilitation sessions, which had the approximate duration of one month.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro SP Gamito, PhD, Study Chair — Universidade Lusófona de Humanidades e Tecnologias; Jorge AG Oliveira, PhD, Principal Investigator — Universidade Lusófona de Humanidades e Tecnologias; Paulo JF Lopes, PhD, Study Director — Universidade Lusófona de Humanidades e Tecnologias
Locations (1):
- Ares do Pinhal. Associação de Recuperação de Toxicodependentes, Sintra, Lisbon District, Portugal

REFERENCES:
- [Derived] Gamito P, Oliveira J, Lopes P, Brito R, Morais D, Silva D, Silva A, Rebelo S, Bastos M, Deus A. Executive functioning in alcoholics following an mHealth cognitive stimulation program: randomized controlled trial. J Med Internet Res. 2014 Apr 17;16(4):e102. doi: 10.2196/jmir.2923. PMID 24742381